CLINICAL TRIAL: NCT04545073
Title: Outcomes of a Trifocal IOL in Post-refractive Patients
Acronym: TrIPLe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vance Thompson Vision ND (Other)
Responsible Party: Sponsor
Other Study IDs: IOL-VTV-01
Record Dates: First submitted 2020-08-21; First posted 2020-09-10 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Post-refractive trifocal IOL
  Interventions: Device: PanOptix

INTERVENTIONS:
Device: PanOptix — Trifocal IOL with ORA in post refractive patients

SUMMARY:
To compare the prediction error of ORA vs formula for post-LASIK cataract patients when PanOptix IOL was implanted. Using post-operative outcomes to determine if preoperative IOL calculations, including Barrett TK, Barrett Universal II, Hill RBF, ASCRS post-refractive calculator, or intraoperative aberrometry is more accurate when the two methods disagree in patients who have had previous refractive surgery undergo cataract surgery.

DETAILED DESCRIPTION:
The study will be non-interventional with data being collected prospectively and retrospectively between at least two surgical sites. All subjects will have previous LASIK and be at least 3 months post op PanOptix implantation. The study will enroll up to 200 patients and a statistical database will be created.

ELIGIBILITY:
Inclusion Criteria:

* Previous myopic refractive surgery
* At least 3 months post op cataract surgery with a trifocal IOL

Exclusion Criteria:

* Pre-existing or subsequent eye condition that interferes with accurate data collection (retinal detachment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Charts from up to 200 myopic post-refractive patients who have received PanOptix will be reviewed at at least two Vance Thompson Vision sites (Fargo, ND and Sioux Falls, SD). All patients will have had ORA used during the cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To determine if preoperative IOL calculations or intraoperative aberrometry is more accurate when the two methods disagree in patients who have had previous refractive surgery undergo cataract surgery. | Pre-op to 9 month visit
  1. Percentage of eyes within +/- .5D of target for each formula and ORA.
  2. Overall % of eyes that have a disagreement between the two methods

SECONDARY OUTCOMES:
Post-operative monocular visual acuity | 3 to 9 month visit
  Monocular Uncorrected Distance, Intermediate, Near Visual Acuity
Post-operative best corrected visual acuity | 3 to 9 month visit
  Manifest refraction, Best Corrected Distance Visual Acuity, Distance Corrected Intermediate, and Near Visual Acuity
Post-operative uncorrected visual acuity | 3 to 9 month visit
  Binocular Uncorrected Distance, Intermediate, Near Visual Acuity, Best Corrected Distance Visual Acuity, Distance Corrected Intermediate, Near Visual Acuity
Post-operative visual acuity | 3 to 9 month visit
  Percentage of eyes with Uncorrected Distance Visual Acuity of 20/20 or better, 20/25 or better, and 20/30 or better
Post-operative visual acuity | 3 to 9 month visit
  Percentage of eyes with Uncorrected Corrected Intermediate Visual Acuity and Distance Corrected Intermediate Visual Acuity 20/20 or better, 20/25 or better, and 20/30 or better
Post-operative visual acuity | 3 to 9 month visit
  Percentage of eyes with Uncorrected Distance Near Visual Acuity and Distance Corrected Near Visual Acuity of 20/20 or better, 20/25 or better, and 20/30 or better
Patient's quality of vision and reported side-effects | 3 to 9 month visit
  Patient satisfaction questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Greenwood, MD, Principal Investigator — Vance Thompson Vision ND
Locations (1):
- Vance Thompson Vision ND, West Fargo, North Dakota, United States